CLINICAL TRIAL: NCT03938038
Title: Guidance of Ultrasound in Intensive Care to Direct Euvolemia: A Cluster Randomized Crossover Comparative Effectiveness Trial (GUIDE Trial)
Brief Title: Guidance of Ultrasound in Intensive Care to Direct Euvolemia
Acronym: GUIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Gabrielle Hatton, Research Fellow, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: HSC-MS-19-0425
Record Dates: First submitted 2019-05-02; First posted 2019-05-06 (Actual); Results first posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-03

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: Randomization will not occur at the individual patient level. Instead, assessment techniques (US-guided versus usual care) will be randomly assigned to care team clusters. Because teams change each month, the assignment will be to US-guided care during the first half or the second half of the month.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Serial ultrasound assessments for GDT, then Usual Care (Active Comparator)
  Interventions: Diagnostic Test: Serial ultrasound assessments for GDT; Diagnostic Test: Usual care
- Usual care, then Serial ultrasound assessments for GDT (Active Comparator)
  Interventions: Diagnostic Test: Serial ultrasound assessments for GDT; Diagnostic Test: Usual care

INTERVENTIONS:
Diagnostic Test: Serial ultrasound assessments for GDT — routine ultrasound assessments of volume status and fluid responsiveness for goal-directed therapy (GDT)-based fluid resuscitation
Diagnostic Test: Usual care — Close hemodynamic cardiac monitoring and volume responsiveness assessment on an unscheduled basis to aid physicians in resuscitation feedback

SUMMARY:
The purpose of this study is to assess the effectiveness of routine ultrasound assessments of volume status and fluid responsiveness for goal-directed therapy (GDT)-based fluid resuscitation in reducing acute kidney injury (AKI) incidence and duration in trauma patients in a teaching institution.

ELIGIBILITY:
Inclusion Criteria:

* Injured patients that are admitted to the trauma ICU

Exclusion Criteria:

* Incarceration
* Pregnancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2020-06-27 (Actual); Study Completion 2020-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabrielle Hatton, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eight different care team clusters will be randomly assigned to either US-guided care or usual care during the 1st half the month and the other technique in the 2nd half. Patient participants will receive either US-guided care or usual care, but not both, and the technique a patient participant receives depends on whether they receive treatment in the 1st or 2nd half of the month. 4 of the 415 enrolled were excluded.
Units Other Than Participants: Care Teams
Period: First Half of the Month (15 Days)
Arm/Group | Serial Ultrasound Assessments for GDT, Then Usual Care | Usual Care, Then Serial Ultrasound Assessments for GDT
Started | 112; 4 Care Teams | 100; 4 Care Teams
Completed | 112; 4 Care Teams | 100; 4 Care Teams
Not Completed | 0; 0 Care Teams | 0; 0 Care Teams
Period: Second Half of the Month (15 Days)
Arm/Group | Serial Ultrasound Assessments for GDT, Then Usual Care | Usual Care, Then Serial Ultrasound Assessments for GDT
Started | 89; 4 Care Teams | 110; 4 Care Teams
Completed | 89; 4 Care Teams | 110; 4 Care Teams
Not Completed | 0; 0 Care Teams | 0; 0 Care Teams

BASELINE CHARACTERISTICS:
Population: Eight different care team clusters will be randomly assigned to either US-guided care or usual care during the 1st half the month and the other technique in the 2nd half. Patient participants will receive either US-guided care or usual care, but not both, and the technique a patient participant receives depends on whether they receive treatment in the 1st or 2nd half of the month. 4 of the 415 enrolled were excluded.
Groups:
- Total: Total of all reporting groups
Arm/Group | Serial Ultrasound Assessments for GDT | Usual Care | Total
Number analyzed (Participants) | 222 | 189 | 411
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 37 [25 to 60] | 39.5 [27 to 60] | 38 [26 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 54 | 130
  Male | 146 | 135 | 281
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44 | 36 | 80
  Not Hispanic or Latino | 151 | 134 | 285
  Unknown or Not Reported | 27 | 19 | 46
Region of Enrollment [Number; unit: participants]
  United States | 222 | 189 | 411

OUTCOME MEASURES:

1. Primary Outcome: Number of Acute Kidney Injury (AKI)-Free Days
Description: AKI will be defined by the Kidney Disease Improving Global Outcomes (KDIGO) criteria, and all stages will be considered AKI:
  Stage 1 - Serum Creatinine 1.5-1.9 times baseline or ≥0.3 mg/dL increase Stage 2 - Serum Creatinine 2-2.9 times baseline Stage 3 - Serum Creatinine 3 times baseline or Increase in serum creatinine to ≥4 mg/dL or Initiation of renal replacement therapy
Time Frame: within 7 days of injury
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Serial Ultrasound Assessments for GDT | Usual Care
Number analyzed (Participants) | 222 | 189
Days | 1 [0 to 2] | 1 [0 to 2]

2. Primary Outcome: Number of Participants Who Receive 3 or More Ultrasound Volume Assessments
Time Frame: within 24 hours of ICU admission
Measure: Count of Participants; unit: Participants
Arm/Group | Serial Ultrasound Assessments for GDT | Usual Care
Number analyzed (Participants) | 222 | 189
Participants | 7 | 0

3. Secondary Outcome: Number of Participants With Acute Kidney Injury (AKI)
Description: as for outcome 1
Time Frame: within the first 7 days of ICU admission
Measure: Count of Participants; unit: Participants
Arm/Group | Serial Ultrasound Assessments for GDT | Usual Care
Number analyzed (Participants) | 222 | 189
Participants | 115 | 119

4. Secondary Outcome: Stage of Acute Kidney Injury (AKI)
Description: as for outcome 1
Time Frame: within the first 7 days of ICU admission
Population: Data were not collected for 107 participants in the Serial Ultrasound Assessments for GDT arm because they did not have AKI. Data were not collected for 70 participants in the usual care arm because they did not have AKI.
Measure: Count of Participants; unit: Participants
Arm/Group | Serial Ultrasound Assessments for GDT | Usual Care
Number analyzed (Participants) | 115 | 119
Participants
  Stage 1 | 67 | 64
  Stage 2 | 32 | 37
  Stage 3 | 16 | 18

5. Secondary Outcome: Number of Participants With Need for Renal Replacement Therapy
Time Frame: within the first 30 days of ICU admission
Measure: Count of Participants; unit: Participants
Arm/Group | Serial Ultrasound Assessments for GDT | Usual Care
Number analyzed (Participants) | 222 | 189
Participants | 16 | 18

6. Secondary Outcome: Quantity of Fluids Administered
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: milliliter (mL)
Arm/Group | Serial Ultrasound Assessments for GDT | Usual Care
Number analyzed (Participants) | 222 | 189
milliliter (mL) | 1562 [489 to 3261] | 1471 [320 to 3428]

7. Secondary Outcome: Quantity of Fluids Administered
Time Frame: 48 hours
Measure: Median (Inter-Quartile Range); unit: milliliter (mL)
Arm/Group | Serial Ultrasound Assessments for GDT | Usual Care
Number analyzed (Participants) | 222 | 189
milliliter (mL) | 1215 [185 to 2938] | 572 [281 to 1408]

8. Secondary Outcome: Type of Fluids Administered
Time Frame: 24 hours
Population: Data were not collected for this outcome measure.
Arm/Group | Serial Ultrasound Assessments for GDT | Usual Care
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Type of Fluids Administered
Time Frame: 48 hours
Population: Data were not collected for this outcome measure.
Arm/Group | Serial Ultrasound Assessments for GDT | Usual Care
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Quantity of Diuretics Administered
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: milliliter (mL)
Arm/Group | Serial Ultrasound Assessments for GDT | Usual Care
Number analyzed (Participants) | 222 | 189
milliliter (mL) | 0 (0) | 0 (0)

11. Secondary Outcome: Quantity of Diuretics Administered
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: milliliter (mL)
Arm/Group | Serial Ultrasound Assessments for GDT | Usual Care
Number analyzed (Participants) | 222 | 189
milliliter (mL) | 0 (0) | 0 (0)

12. Secondary Outcome: Time to Lactate Normalization
Time Frame: within the first 7 days of ICU admission
Population: Data were not collected for this outcome measure.
Arm/Group | Serial Ultrasound Assessments for GDT | Usual Care
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Time to Creatinine Concentration <1.5 mg/dL or to Prehospital Baseline
Time Frame: within the first 7 days of ICU admission
Population: Data were not collected for this outcome measure.
Arm/Group | Serial Ultrasound Assessments for GDT | Usual Care
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Time to Base Excess Normalization
Time Frame: within the first 7 days of ICU admission
Population: Data were not collected for this outcome measure.
Arm/Group | Serial Ultrasound Assessments for GDT | Usual Care
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Number of Ventilator-free Days
Time Frame: within first 30 days after injury
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Serial Ultrasound Assessments for GDT | Usual Care
Number analyzed (Participants) | 222 | 189
days | 29 [26 to 30] | 29 [26 to 30]

16. Secondary Outcome: Number of ICU-free Days
Time Frame: within first 30 days after injury
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Serial Ultrasound Assessments for GDT | Usual Care
Number analyzed (Participants) | 222 | 189
days | 26 [22 to 28] | 26 [22 to 28]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Serial Ultrasound Assessments for GDT | Usual Care
All-Cause Mortality (participants affected / at risk) | 21/222 | 15/189
Serious Adverse Events (participants affected / at risk) | 23/222 | 15/189
Other Adverse Events (participants affected / at risk) | 115/222 | 119/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Serial Ultrasound Assessments for GDT (N=222) | Usual Care (N=189)
Death (General disorders) | 21 (21) | 15 (15)
New Onset Congestive Heart Failure (Cardiac disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Serial Ultrasound Assessments for GDT (N=222) | Usual Care (N=189)
Acute Kidney Injury (Renal and urinary disorders) | 115 | 119

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-03): https://cdn.clinicaltrials.gov/large-docs/38/NCT03938038/Prot_SAP_000.pdf